CLINICAL TRIAL: NCT04807335
Title: Bioavailability Study of Intranasal CT001 in Healthy Volunteers
Brief Title: Study of CT001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cessatech A/S (Industry)
Collaborators: Dantrials Aps (Industry); Smerud Medical Research International AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PDC 01-0204
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Bioavailability
MeSH Terms: interventions — Ketamine; Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational medicinal product CT001 (Experimental): intranasal dosage of CT001
  Interventions: Drug: CT001
- Comparator 1 (Active Comparator): Ketamine 10mg iv
  Interventions: Drug: Ketamine
- Comparator 2 (Active Comparator): Sufentanil 10mcg iv
  Interventions: Drug: sufentanil

INTERVENTIONS:
Drug: CT001 — nasal spray
  Arms: Investigational medicinal product CT001
Drug: Ketamine — iv single dose
  Arms: Comparator 1
Drug: sufentanil — iv single dose
  Arms: Comparator 2

SUMMARY:
A phase 1, three arms, cross over comparison study to evaluate bioavailability, pharmacokinetics and safety of intra nasal CT001 in healthy volunteers.

DETAILED DESCRIPTION:
A single site phase 1 study including a randomised, open label, three periods, single dose, cross over design in 12 healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 up to 55 years
* Non-smokers
* Body mass index (BMI) from 18.5 kg/m2 up to 30 kg/m2 v) Categorized as American Society of Anesthesiologists (ASA)
* Physical Status Class 1 or 2
* Clinically normal medical history, physical findings, vital signs, ECG and laboratory values.

Exclusion Criteria:

* Mental illness
* Opioid Risk Tool score of >3
* Pain Catastrophizing Scale score, total points >30
* Hospital Anxiety and Depression Scale (HADS), points ≥11 for anxiety or ≥11 points for depression
* Daily intake of analgesics
* History of alcohol or drug abuse or use of illicit drugs.
* Use of prescription drugs within 14 days or over-the-counter drugs 24 hours (intranasal medication 48 hours) prior to the first dose of study medication.
* Participant showing abnormal nasal cavity/airway
* History or presence of allergy to the study drug or drugs of this class, or a history of drug or other allergy.
* Positive tests for HIV, hepatitis B and hepatitis C
* Positive COVID-19 test or clinical symptoms of COVID-19
* Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 30 days of signing the informed consent for this trial
* Blood donation within 4 weeks prior to the first dosing visit

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
concentration of CT001 in the blood | baseline, 3, 5, 10, 15, 30, 60, 90, 180, 240 minutes and 6, 9, 24, 32, 48 hours after dose
  maximum concentration over time C(max),
Total amount of CT001 in the blood over time | baseline, 3, 5, 10, 15, 30, 60, 90, 180, 240 minutes and 6, 9, 24, 32, 48 hours after dose
  Area under the curve calculated from t=0 to t= 48 hours

SECONDARY OUTCOMES:
distribution and elimination of CT001 | baseline, 3, 5, 10, 15, 30, 60, 90, 180, 240 minutes and 6, 9, 24, 32, 48 hours after dose
  Volume of distribution
number of study participants with adverse events | from baseline to 48 hours post dose
  Number andproportion of adverse events,
elimination of CT001 | from baseline to 48 hours
  Half time
vital signs | from baseline to 48 hours
  heart rate, blood pressure, respiratory rate and blood oxygen level

CONTACTS AND LOCATIONS:
Overall Officials: Mads Werner, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Dantrials, Copenhagen, DK, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: sponsor's homepage — http://cessatech.com